CLINICAL TRIAL: NCT04971603
Title: The Effectiveness and Safety of Acupuncture for Elderly Patients of Stroke: a Pragmatic Study of Acupuncture for Primary Care
Brief Title: The Effectiveness and Safety of Acupuncture for Elderly Patients of Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acupuncture for stroke
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-01

CONDITIONS: Stroke
Keywords: Stroke; Chinese Medicine; Acupuncture
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: This is a single arm prospective study. A total of 500 eligible patients will be recruited for 24-week treatment and 12-week follow up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture treatment group (Experimental): The patients will receive 24-week acupuncture treatment and 12-week follow up. Seven visits will be arranged within the 24-wk treatment period and at the end of study at wk 6, 10, 14, 18, 22, 26 and 38 for medical consultation and investigation.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — All acupuncture operations were done by registered Chinese medicine practitioner. Sterile, disposable acupuncture needles (0.25mmin diameter and 40mmin length) were used, which were purchased from HuaTuo acupuncture instrument.
  Principal points: Neiguan (PC 6) *, Sanyinjia (SP 6) *, Weizhong (BL 40) *, Baihui (GV 20), Shuigou (GV 26) *, Zusanli (ST 36) *, Quchi (LI 11) *, Waiguan (TE 5) *, Hegu (LI 4) *, Huantiao (GB 30) *, Yanglingquan (GB 34)* (Grading of recommendation: C, level of evidence: IV).
  Supplementary points: If upper limbs hemiplegia occurs, add Jianliao (TE 14) and Shousanli (LI 10); if lower limbs hemiplegia occurs, add Xuanzhong (GB 39) and Taichong (LR 3); if a deviation of the mouth or tongue occurs, add Dicang (ST 4) and Jiache (ST 6).

SUMMARY:
Stroke and its sequelae are a major indication for acupuncture. The specific aims of this study are to assess the feasibility of pragmatic clinical trial on acupuncture in primary care setting and evaluate the effectiveness and safety of acupuncture for stroke rehabilitation in Hong Kong.

DETAILED DESCRIPTION:
The study will help to develop ap treatment patterns for stroke rehabilitation of elderly patients in Hong Kong. The specific aims of this study are to assess the feasibility of pragmatic clinical trial on acupuncture in primary care setting and evaluate the effectiveness and safety of acupuncture for stroke rehabilitation on motor, sensation, speech, swallowing, cognitive, and other neurological functions.

This study includs 2-week run-in, 24-week treatment, 12-week follow up and 9 visits at week 0, 2, 6, 10, 14, 18, 22, 26 and 38. The investigator will recruit totally 500 patients fulfiling the eligibility criteria in four neighbourhood elderly centres of The Hong Kong Sheng Kung Hui Welfare Council and Chinese medicine clinics of Hong Kong Baptist University. Acupuncture treatment will be applied to the patients and seven visits will be arranged within the 24-wk treatment period providing medical consultation and recording improvement and any adverse effect.

ELIGIBILITY:
Inclusion Criteria:

- Participants who meet the following criteria will be included: (1) 35~90 years or older; (2) discharged from hospital; (3) diagnosed with cerebral hemorrhage or cerebral infarction through brain computed tomography (CT) or magnetic resonance imaging (MRI); (4) stable vital signs; and (5) voluntary participation with informed consents signed in this study.

Exclusion Criteria:

- The following participants are excluded: (1) patients with unconsciousness, aphasia, and cognitive dysfunction (Mini-Mental State Examination-Korean version (MMSE-K) <24); (2) those with a past history of brain disease (e.g., mental illness, consciousness disorder due to head trauma, previous brain surgery, or spastic disease); (3) those with severe heart, liver, or kidney disease or bleeding disorders; (4) those with other serious diseases (e.g., cancer, dementia (Alzheimer's disease or dementia of Lewy body), Parkinson's disease, and Parkinson's syndrome); (5) those who participated in other clinical trials within last three months; (6) those with needle phobia; and (7) pregnant or lactating female patients.

Ages: 35 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Activities of daily living (ADL) scores | 9 months
  ADL is commonly utilized to indicate the patient's functioning condition and level of care assistance by the Hospital Authority in Hong Kong.

SECONDARY OUTCOMES:
Mini-mental state examination (MMSE) | 9 months
  The MMSE test is a standard tool for cognitive assessment in the clinical setting. It is a 10-minute bedside measure of impaired thinking in undeveloped, uneducated, diseased, or very old populations. The summed score of the individual items indicates the current severity of cognitive impairment.
Traditional Chinese Medicine Syndrome Score Scale (TCMSSS) | 9 months
  The TCMSSS is based on <Criteria for diagnosis and curative effect evaluation of stroke>. Total scores range from 0 to 52, with scores above 40 indicating very severe neurological impairment, scores of 14 to 39 suggesting moderately severe to severe impairment, and scores below 13 indicating mild impairment.
Constitution in Chinese Medicine Questionnaire (CCMQ) | 9 months
  The CCMQ is applied to evaluate body constitution of each patient by score (Balanced Constitution, Qi-deficient Constitution, Yang-deficient Constitution, Yin-deficient Constitution, Phlegm-dampness Constitution, Damp-heat Constitution, Stagnant Blood Constitution, Stagnant Qi Constitution, and Inherited Special Constitution).

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong, Kowloon Tong, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided